CLINICAL TRIAL: NCT06770855
Title: A Phase II Study of Total Consolidative Metastasis-and-primary Directed Therapy (MPDT) for Renal Cell Carcinoma (RCC).
Brief Title: Consolidative Metastasis and Primary Directed Therapy (MPDT) for Renal Cell Carcinoma (RCC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 33824; IRB#857362 (Other: [University of Pennsylvania IRB)
Record Dates: First submitted 2024-12-23; First posted 2025-01-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Total consolidative MPDT (Experimental): Participants will discontinue systemic anti-cancer therapy for metastatic RCC, and standard of care definitive procedures or metastatic RCC. These procedures include one or more of the following: surgery (e.g. nephrectomy, metastasectomy, lymph node dissection), percutaneous cryoablation and/or radiotherapy (SAbR or other definitive radiotherapy).
  Interventions: Procedure: Total consolidative MPDT

INTERVENTIONS:
Procedure: Total consolidative MPDT — After stopping systemic anti-cancer therapy for metastatic RCC, participant will receive one or more of the following: surgery (e.g. nephrectomy, metastasectomy, lymph node dissection), percutaneous cryoablation and/or radiotherapy (SAbR or other definitive radiotherapy).

SUMMARY:
This is a non-randomized, open-label phase II study designed to estimate 12-month treatment-free survival rate following total consolidative metastasis-and-primary directed therapy (MPDT) among patients with partial response/stable disease after at least 6 months of immune checkpoint blockade-based therapy for metastatic clear cell RCC. The investigators hypothesize that patients who undergo total consolidative MPDT followed by systemic therapy discontinuation will have a 12-month treatment-free survival rate of 32% compared to a null hypothesis of 13%

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of clear cell renal cell carcinoma (mixed histology acceptable but must have clear cell component)
* Metastatic clear cell RCC with 5 or fewer metastases at enrollment (excluding pulmonary nodules <1.0cm)
* Stable disease or partial response as assessed by investigators following at least 6 months of immune checkpoint blockade-based therapy.
* Has disease amenable for total consolidative focal therapy (this will be determined by a multidisciplinary team which may include a combination of medical oncologists, urologists, interventional radiologists, and radiation oncologists).
* ECOG performance status < 2
* Must have archival tissue (slide or Formalin-Fixed Paraffin-Embedded tissue) preceding prior systemic treatment for comparison to tissue from consolidation
* Consolidation surgery and biopsies are strongly encouraged to be within 42 days +/- 7 days of holding systemic therapy.

Exclusion Criteria:

* Subjects who have progressed during the first 6 months of immune checkpoint-blockade based therapy as determined by study investigator.
* Subjects who have a need for urgent focally directed therapy (i.e. symptomatic brain or spinal metastases). Stable spinal metastases resected and/or treated with SBRT in advance of or concurrently with immune checkpoint-blockade based therapy are allowed to participate.
* Any female of child-bearing potential who has a positive urine pregnancy test within 72 hours before screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Participants must be excluded/discontinued from the trial in the event of a positive or borderline positive serum pregnancy test result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-04-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-free survival | From discontinuation of anti-cancer therapy until resumption of systemic therapy, first date of additional focally-directed therapy or death, whichever comes first, assessed up to 60 months.
  Treatment-free survival, defined as the time from discontinuation of anti-cancer therapy until either: 1) the resumption of systemic therapy; 2) the first date of additional focally-directed therapy; or 3) death.

SECONDARY OUTCOMES:
Recurrence-free survival | From completion of total consolidative MPDT until investigator-assessed disease recurrence, assessed up to 60 months..
  Recurrence-free survival, defined as the time from completion of total consolidative MPDT until investigator-assessed disease recurrence.
Grade 3 or higher adverse events | From completion of total consolidative MPDT until investigator-assessed disease recurrence, assessed up to 60 months.
  Grade 3 or higher adverse events according to the Clavien-Dindo scale (surgery), Society for Interventional Radiology scale (percutaneous cryoablation), or the CTCAE v5.0 (radiotherapy)

OTHER OUTCOMES:
Identify an immune signature that correlates with treatment free survival | At week 6 and week 12 following systemic therapy initiation, at the time of study enrollment and following total consolidative MPDT, through study completion, estimated to be 36 months.
  The investigators will broadly interrogate immune cell types from the peripheral blood and tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Haas, MD, Principal Investigator — Penn Medicine
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States